CLINICAL TRIAL: NCT01014000
Title: OPTimization of Left-Ventricular Lead Implantation by Echocardiography- E-OPT Study
Brief Title: Comparative Study to Examine Whether Echocardiography Performed During Cardiac Resynchronization Therapy Device Implantation Can Improve the Response Rate
Acronym: E-OPT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: On reviewing of new data
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Ngai Yin Chan, Dr, Princess Margaret Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EOPT01
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy; Echocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empirical (Active Comparator): Empirical implantation of the left ventricular lead during cardiac resynchronization therapy device implantation
  Interventions: Device: Empirical group
- Echocardiography-guided approach (Experimental): Echocardiography-guided implantation of the left ventricular lead during cardiac resynchronization therapy device implantation
  Interventions: Device: Echocardiography-guided approach

INTERVENTIONS:
Device: Empirical group — Empirical implantation of the left ventricular lead during cardiac resynchronization therapy device implantation
  Arms: Empirical
Device: Echocardiography-guided approach — Echocardiography-guided implantation of the left ventricular lead during cardiac resynchronization therapy device implantation
  Arms: Echocardiography-guided approach

SUMMARY:
Empirical implantation of the left ventricular lead is the prevailing practice in cardiac resynchronization therapy device implantation. The response rate to the therapy has been uniformly 70% only despite various methods to screen patients before device implantation. This study tested the hypothesis that echocardiography to assess acute resynchronization of the left ventricle during device implantation may improve the response rate to the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SR or AF, indicated for CRT procedures (NYHA Class III or ambulatory Class IV despite optimal medical therapy, QRSd≥120ms and LVEF≤35%)
2. Patients with ischaemic or non-ischaemic cardiomyopathy can be recruited

Exclusion Criteria:

1. Patients already implanted with an implantable cardiac device, undergoing device upgrade or generator replacement
2. Patients who aged less than 18 or over 80.
3. Patients who are pregnant.
4. Patients who cannot give informed consent.
5. Patients who are judged to have severe mental impairment and cannot report symptoms of heart failure during follow-up.
6. Patients who have comorbid congenital heart disease.
7. Patients who have severe valvular heart disease, apart from severe mitral regurgitation.
8. Patients who have unstable angina or who are within 1 month of myocardial infarction.
9. Patients who have severe lung disease and accurate clinical assessment for heart failure symptoms cannot be performed.
10. Patients who have poor echocardiographic windows precluding reliable echocardiographic examination during baseline assessment, CRT procedures or follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Clinical response (Improvement in functional class status by at least one NYHA Class or ≥10% increase in 6-minute hall walk distance) to CRT | 6 months after device implantation

SECONDARY OUTCOMES:
Echocardiographic response of ≥15% reduction in LVESV | 6 months after device implantation
Echocardiographic response of absolute increase of ≥5% in LVEF | 6 months after device implantation
Biochemical response with reduction of BNP level≥15% | 6 months after device implantation

CONTACTS AND LOCATIONS:
Overall Officials: Ngai Yin Chan, MBBS, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Hong Kong, China